CLINICAL TRIAL: NCT00785187
Title: Randomized Open Crossover Study Researching Affect of Dose Rate on UVR Induced Skin Erythema
Brief Title: Affect of Dose Rate on UVR Induced Skin Erythema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Goldenhersh, Michael, M.D. (Individual)
Responsible Party: Dr. Michael Goldenhersh, Dr. Goldenhersh's Dermatology Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: goldenhersh1
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-11

CONDITIONS: Erythema
Keywords: UVB induced skin erythema
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: exposure to UVB radiation — exposure to UVB radiation for limited time in order to establish subject's minimal erythema dose.

SUMMARY:
Purpose of study: Evaluation of the affect of dose rate on UVR induced skin erythema.

Study design: A single-center, prospective, randomized, crossover, open study.

Number of patients: 20-40

Patient population: Healthy volunteers

Control: Different sites on patients body

Procedure duration: Total 3-5 hours (4 visits)

Duration of follow up: 4 days

Duration of study: Up to 6 months

Primary objectives: To examine the difference in erythemal response as a function of dose rate, and to assess the total amount of energy that is theoretically transmitted through a sunscreen within the range of SPF 2-10.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin types I-III.
* Age 18-60.
* Absence of obvious sun damage on the volar side of the forearm or other exposure sites.
* Absence of exposure of the arms or other exposure sites to sunlight for two weeks prior to the experiment.

Exclusion Criteria:

* History of skin cancer.
* Multiple nevi or atypical nevi on the forearm.
* Signs of sun damage on the volar side of the forearm or other exposure sites.
* Mentally incompetent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
To examine the difference in erythemal response as a function of dose rate, and to assess the total amount of energy that is theoretically transmitted through a sunscreen within the range of SPF 2-10 | end of study